CLINICAL TRIAL: NCT02476630
Title: Thenar Tissue Oxygen Concentration (StO2): A Non-invasive Surrogate for Central Venous Oxygen Saturation (ScvO2)
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201500482
Record Dates: First submitted 2015-06-12; First posted 2015-06-19 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Oxygen Concentration Levels
MeSH Terms: interventions — Blood Gas Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study subjects: All participants will have a measurement of the tissue oxygen concentration (StO2) level after applying the noninvasive probe to the thenar eminence. This measurement is done at the same time as blood gases(ScvO2) from the central venous catheter is obtained. The StO2 measurement is documented once for the subject in the study.
  Interventions: Device: StO2 measurement; Other: Blood Gases

INTERVENTIONS:
Device: StO2 measurement — All participants will have a measurement of the tissue oxygen concentration (StO2) level after applying the noninvasive probe to the thenar eminence. This measurement is done at the same time as a blood gas from the central venous catheter is obtained. The StO2 measurement is documented once for the subject in the study.
  Other Names: InSpectraTM StO2 monitor
Other: Blood Gases — All participants will have a measurement of the tissue oxygen concentration (StO2) level after applying the noninvasive probe to the thenar eminence. This measurement is done at the same time as a blood gas from the central venous catheter is obtained. The StO2 measurement is documented once for the subject in the study.
  Other Names: central venous oxygen saturation (ScvO2)

SUMMARY:
Oxygen concentration for patients undergoing cardiac catheterization and during admission to an intensive care unit is important outcome measure for clinical care. Currently, the tool used to monitor the oxygen concentration is a central venous access positioned in the superior vena cava or in the pulmonary artery to monitor the central venous oxygen saturation (ScvO2). However, it is invasive and not always possible due to a lack of a central line access. In this research study, the investigator would like use a noninvasive means for the ScvO2 by using the thenar tissue oxygen concentration (StO2). The primary aim for the study is to determine if the thenar StO2 correlates with ScvO2 and can serve as a noninvasive surrogate for ScvO2.

DETAILED DESCRIPTION:
Participants will be undergoing a cardiac catheterization at Shands Children's Hospital or will be admitted to the intensive care unit, and as part of the clinical care either a central venous access positioned in the superior vena cava or in the pulmonary artery. As a part of the routine clinical care blood gases are frequently taken for continuous evaluation of therapy to monitor the central venous oxygen saturation (ScvO2). A measurement of thenar tissue oxygen concentration will be timed with a central venous blood gas draw to monitor the tissue oxygen concentration (StO2).

The StO2 measurement will be taken by using the InSpectraTM StO2 monitor manufactured by Hutchinson Technology Inc. after applying the noninvasive clip on probe to the thenar eminence of the right hand to measure the StO2 level. After a stable reading is obtained for 60 seconds it will be recorded.

The two different measurements of oxygen concentration will be compared to determine if a correlation exists.

ELIGIBILITY:
Inclusion Criteria:

1. Age 1 month to 21 years of age admitted to the intensive care unit or undergo cardiac catheterization at Shands Children's Hospital and have a central venous access positioned in the superior vena cava or pulmonary artery.

Exclusion Criteria:

1. Age less than 1 month or more than 21 years
2. Burns of the hand
3. Infection of hand
4. Fracture of upper extremity
5. Hematoma of hand over thenar eminence

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be undergoing a cardiac catheterization atan area Children's Hospital or will be admitted to the intensive care unit, and as part of the clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Measurement of tissue oxygen concentration (StO2) percentage | Day 1
  The use of the InSpectraTM StO2 monitor manufactured by Hutchinson Technology INC. will be used to measure the StO2 level after applying the noninvasive probe to the thenar eminence.

SECONDARY OUTCOMES:
Comparison of thenar StO2 oxygen saturation calculations between central venous oxygen saturation (ScvO2) calculations. | Day 1
  The correlation between StO2 and ScvO2 will be determined by using Pearson's correlation test.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Samraj, MD, Principal Investigator — University of Florida , Gainesville, Florida, United States, 32610
Locations (1):
- Shands Childrens Hospital UF Health, Gainesville, Florida, United States

REFERENCES:
- [Background] Crookes BA, Cohn SM, Bloch S, Amortegui J, Manning R, Li P, Proctor MS, Hallal A, Blackbourne LH, Benjamin R, Soffer D, Habib F, Schulman CI, Duncan R, Proctor KG. Can near-infrared spectroscopy identify the severity of shock in trauma patients? J Trauma. 2005 Apr;58(4):806-13; discussion 813-6. doi: 10.1097/01.ta.0000158269.68409.1c. PMID 15824660
- [Background] Beilman GJ, Groehler KE, Lazaron V, Ortner JP. Near-infrared spectroscopy measurement of regional tissue oxyhemoglobin saturation during hemorrhagic shock. Shock. 1999 Sep;12(3):196-200. doi: 10.1097/00024382-199909000-00005. PMID 10485597
- [Background] Taylor DE, Simonson SG. Use of near-infrared spectroscopy to monitor tissue oxygenation. New Horiz. 1996 Nov;4(4):420-5. PMID 8968975
- [Background] Mesquida J, Masip J, Gili G, Artigas A, Baigorri F. Thenar oxygen saturation measured by near infrared spectroscopy as a noninvasive predictor of low central venous oxygen saturation in septic patients. Intensive Care Med. 2009 Jun;35(6):1106-9. doi: 10.1007/s00134-009-1410-y. Epub 2009 Jan 29. PMID 19183952